CLINICAL TRIAL: NCT06706323
Title: Predictive Modelling of Clinically Significant Depressive Symptoms After Coronary Artery Bypass Graft Surgery
Brief Title: Depressive Symptoms After Cardiac Surgery
Acronym: PCD
Status: Recruiting | Type: Observational
Sponsor: Roland von Känel (Other)
Collaborators: Triemli Hospital (Other); ETH Zurich (Other); University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Roland von Känel, Prof. Dr. med., University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: BASEC 2023-02040; 215033 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases; Coronary Artery Disease; Heart Diseases; Depression; Depressive Symptoms; Anxiety; Posttraumatic Stress Disorder; Quality of Life; Psychological Well-Being; Postoperative Complications
Keywords: Coronary Artery Bypass Graft; Coronary Artery Bypass Grafting; Coronary Artery Bypass Surgery; CABG; Inflammation; Interoception; Clinically Significant Depressive Symptoms; CSDS; Patient Health Questionnaire-9; PHQ-9; Postoperative Depression; Algorithms; Prediction; Predictive Modeling; Machine Learning
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Heart Diseases; Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Psychological Well-Being; Postoperative Complications; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training group: From the final cohort of 300 participants, 200 will be recruited at Hospital I (University Hospital Zurich) to form the training group for developing the optimal statistical model.
- Test group: From the final cohort of 300 participants, the remaining 100 will be recruited at Hospital II (Stadtspital Zurich Triemli) to form the test group for validating the final model.

SUMMARY:
The primary goal of this project is to develop a predictive model for clinically significant depressive symptoms (CSDS) in patients undergoing coronary artery bypass graft (CABG) surgery, using pre- and perioperative data. CSDS occur in about 30 percent of CABG patients, which is four times higher than in the general population. These symptoms are linked to poor quality of life and increased morbidity and mortality. The aim is to create a model that can identify patients at risk for postoperative depression. This tool could help clinicians make informed decisions and take preventive measures to manage depression after surgery.

DETAILED DESCRIPTION:
In patients undergoing coronary artery bypass graft (CABG) surgery, the prevalence of clinically significant depressive symptoms (CSDS) is about 30 percent, four times higher than the 12-month prevalence in the general population. CSDS are associated with poor quality of life and increased morbidity and mortality. While several predictors of post-CABG CSDS have been identified, no prognostic model exists.

The aim of this project is to develop a predictive model for post-surgery CSDS in CABG patients using pre- and perioperative data. A prognostic prediction model for CSDS 6 weeks post-CABG, will be developed using demographic, psychometric, medical, inflammation, and cardiac interoception data. Machine learning algorithms will be employed for data analysis. A cohort of 350 participants from two hospitals will be recruited, with 300 participants expected to complete the study. Data will be divided into training (200 participants) and testing (100 participants) sets. Nested cross-validation will prevent overfitting. Both binary and regression prediction models will be used. Additionally, a simpler model will be developed to increase generalizability.

The prediction model will identify CABG patients at risk of post-surgery CSDS. The model will help identify patients at risk for CSDS before surgery, enabling early interventions. Clinicians can make precision medicine decisions to prevent or manage CSDS, improving postoperative psychological well-being. Additionally, the study could advance understanding of the mechanisms linking depression and coronary heart disease, particularly in relation to inflammation and interoception.

ELIGIBILITY:
Inclusion Criteria:

* Elective Off-Pump CABG or CABG, either isolated or combined with valve intervention
* Men and women, aged between 18 and 90 years
* Sufficient knowledge of German language in reading and understanding
* Oral and Signed consent form
* Ability and Willingness to follow the study protocol

Exclusion Criteria:

* Cognitive impairment according to a score of ≤ 7 (maximum score = 9) on a modified version of a short version of the Mini-Mental State Examination and the Brief Interview for Mental Status
* Any serious comorbid non-cardiac medical condition likely to cause death within 1 year (e.g. metastatic cancer)
* Active psychotic symptoms (assessed with two items from the Youth Psychosis At Risk Questionnaire), substance abuse and/or dependence within the past 6 months (assessed with a single-item questionnaire), and/or active suicidal ideations (assessed with a single item from the M.I.N.I.).
* Acute or emergency CABG

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include 300 patients undergoing coronary artery bypass graft (CABG) surgery, recruited from two hospitals: the University Hospital Zurich (USZ) and the Municipal Hospital of Zurich - Triemli. Of these, 200 patients will be in the training group and 100 in the test group for developing and validating a predictive model for post-surgery depressive symptoms. Participants will be recruited consecutively, with inclusive criteria regarding sex and an upper age limit of 90 years to enhance eligibility and generalizability. As no literature suggests differences in depressive symptoms based on surgery type, patients will be included regardless of whether their CABG is isolated or combined with valve intervention.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) score ≥10 (yes/no) at 6 weeks post-CABG | Baseline (1 day before CABG surgery) and Follow Up (6 weeks after CABG surgery)
  The Patient Health Questionnaire (PHQ)-9 will assess the severity of self-rated depressive symptoms over the last two weeks. It covers the nine Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5) criteria for major depression, with symptoms rated on a 4-point Likert scale. Scores range from 0 to 27, with higher scores indicating more severe symptoms. A score of 10 or higher corresponds to a diagnosis of depression, with 88 percent sensitivity and specificity.
  As the best cut-off for post-CABG CSDS is difficult to determine a priori for a prediction model, a two complementary approaches for the analysis will be used, correcting for multiple tests when assessing the significance of the accuracy of the prediction model. One approach frames the prediction challenge as a binary classification problem and uses a PHQ-9 cut-off score ≥10 for defining the presence versus absence of CSDS.

SECONDARY OUTCOMES:
PHQ-9 score continuous at 6 weeks post-CABG | Baseline (1 day before CABG surgery) and Follow Up (6 weeks after CABG surgery)
  The PHQ-9 will assess the severity of self-rated depressive symptoms over the last two weeks. It covers the nine DSM-5 criteria for major depression, with symptoms rated on a 4-point Likert scale. Scores range from 0 to 27, with higher scores indicating more severe symptoms. A score of 10 or higher corresponds to a diagnosis of depression, with 88 percent sensitivity and specificity.
  As the best cut-off for post-CABG CSDS is difficult to determine a priori for a prediction model, a two complementary approaches for the analysis will be used, correcting for multiple tests when assessing the significance of the accuracy of the prediction model. The second approach views the prediction challenge as a regression problem and tries to predict individual PHQ-9 scores without applying any threshold.
General Anxiety Disorder (GAD-7) score ≥10 (yes/no) at 6 weeks post-CABG | Baseline (1 day before CABG surgery) and Follow Up (6 weeks after CABG surgery)
  The General Anxiety Disorder (GAD)-7 questionnaire will assess self-rated anxiety symptoms over the past two weeks. Seven items are rated on a 4-point Likert scale, with total scores ranging from 0 to 21. A score of 10 or higher indicates moderate to severe anxiety, corresponding to a GAD diagnosis with 89% sensitivity and 82% specificity.
  As the best cut-off for post-CABG GAD is difficult to determine a priori for a prediction model, a two complementary approaches for the analysis will be used, correcting for multiple tests when assessing the significance of the accuracy of the prediction model. One approach frames the prediction challenge as a binary classification problem and uses a GAD-7 cut-off score ≥10 for defining the presence versus absence of GAD.
GAD-7 score continuous at 6 weeks post-CABG | Baseline (1 day before CABG surgery) and Follow Up (6 weeks after CABG surgery)
  The GAD-7 questionnaire will assess self-rated anxiety symptoms over the past two weeks. Seven items are rated on a 4-point Likert scale, with total scores ranging from 0 to 21. A score of 10 or higher indicates moderate to severe anxiety, corresponding to a GAD diagnosis with 89% sensitivity and 82% specificity.
  As the best cut-off for post-CABG GAD is difficult to determine a priori for a prediction model, a two complementary approaches for the analysis will be used, correcting for multiple tests when assessing the significance of the accuracy of the prediction model. The second approach views the prediction challenge as a regression problem and tries to predict individual GAD-7 scores without applying any threshold.
PTSD (Post-traumatic Stress Disorder) Checklist for DSM-5 (PCL-5) score ≥33 at 6 weeks post-CABG | Baseline (1 day before CABG surgery) and Follow Up (6 weeks after CABG surgery)
  The PTSD Checklist for DSM-5 (PCL-5) will assess CABG surgery-induced posttraumatic stress. It is a 20-item self-report measure evaluating the DSM-5 PTSD symptoms over the past month. Items are rated on a 5-point Likert scale, with scores of 33 or higher indicating probable PTSD.
  As the best cut-off for post-CABG PTSD is difficult to determine a priori for a prediction model, a two complementary approaches for the analysis will be used, correcting for multiple tests when assessing the significance of the accuracy of the prediction model. One approach frames the prediction challenge as a binary classification problem and uses a PCL-5 cut-off score ≥33 for defining the presence versus absence of PTSD.
PCL-5 score continuous at 6 weeks post-CABG | Baseline (1 day before CABG surgery) and Follow Up (6 weeks after CABG surgery)
  The PCL-5 will assess CABG surgery-induced posttraumatic stress. It is a 20-item self-report measure evaluating the DSM-5 PTSD symptoms over the past month. Items are rated on a 5-point Likert scale, with scores of 33 or higher indicating probable PTSD.
  As the best cut-off for post-CABG PTSD is difficult to determine a priori for a prediction model, a two complementary approaches for the analysis will be used, correcting for multiple tests when assessing the significance of the accuracy of the prediction model. The second approach views the prediction challenge as a regression problem and tries to predict individual PCL-5 scores without applying any threshold.
Short-Form Health Survey-12 (SF-12) mental health component score at 6 weeks post-CABG | Baseline (1 day before CABG surgery) and Follow Up (6 weeks after CABG surgery)
  The Short-Form Health Survey (SF-12) will assess physical and mental health-related quality of life (QoL) over the last four weeks, covering aspects such as physical functioning, pain, vitality, social functioning, and mental health.
SF-12 physical health component score at 6 weeks post-CABG | Baseline (1 day before CABG surgery) and Follow Up (6 weeks after CABG surgery)
  The SF-12 will assess physical and mental health-related quality of life (QoL) over the last four weeks, covering aspects such as physical functioning, pain, vitality, social functioning, and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Omer Dzemali, Prof. Dr., Principal Investigator — Stadtspital Zürich Triemli, Klinik für Herzchirurgie, Birmensdorferstr. 497, 8063 Zurich, Switzerland; Roland v Känel, Prof. Dr., Principal Investigator — University Hospital Zurich, Dept. of Consultation-Liaison Psychiatry, Haldenbachstr. 16/18, 8091 Zurich, Switzerland
Locations (2):
- Switzerland (2):
  - Stadtspital Zürich (City Hospital Zurich) Triemli, Zurich
  - University Hospital Zurich (USZ), Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chocron S, Vandel P, Durst C, Laluc F, Kaili D, Chocron M, Etievent JP. Antidepressant therapy in patients undergoing coronary artery bypass grafting: the MOTIV-CABG trial. Ann Thorac Surg. 2013 May;95(5):1609-18. doi: 10.1016/j.athoracsur.2013.02.035. Epub 2013 Apr 6. PMID 23566649
- [Background] Correa-Rodriguez M, Abu Ejheisheh M, Suleiman-Martos N, Membrive-Jimenez MJ, Velando-Soriano A, Schmidt-RioValle J, Gomez-Urquiza JL. Prevalence of Depression in Coronary Artery Bypass Surgery: A Systematic Review and Meta-Analysis. J Clin Med. 2020 Mar 26;9(4):909. doi: 10.3390/jcm9040909. PMID 32225052
- [Background] Guo P. Preoperative education interventions to reduce anxiety and improve recovery among cardiac surgery patients: a review of randomised controlled trials. J Clin Nurs. 2015 Jan;24(1-2):34-46. doi: 10.1111/jocn.12618. Epub 2014 Jun 3. PMID 24894181
- [Background] Protogerou C, Fleeman N, Dwan K, Richardson M, Dundar Y, Hagger MS. Moderators of the effect of psychological interventions on depression and anxiety in cardiac surgery patients: A systematic review and meta-analysis. Behav Res Ther. 2015 Oct;73:151-64. doi: 10.1016/j.brat.2015.08.004. Epub 2015 Aug 14. PMID 26319588
- [Background] Ravven S, Bader C, Azar A, Rudolph JL. Depressive symptoms after CABG surgery: a meta-analysis. Harv Rev Psychiatry. 2013 Mar-Apr;21(2):59-69. doi: 10.1097/HRP.0b013e31828a3612. PMID 23656830
- [Background] Takagi H, Ando T, Umemoto T; ALICE (All-Literature Investigation of Cardiovascular Evidence) Group. Perioperative depression or anxiety and postoperative mortality in cardiac surgery: a systematic review and meta-analysis. Heart Vessels. 2017 Dec;32(12):1458-1468. doi: 10.1007/s00380-017-1022-3. Epub 2017 Jul 13. PMID 28702898
- [Background] Tully PJ, Baker RA. Depression, anxiety, and cardiac morbidity outcomes after coronary artery bypass surgery: a contemporary and practical review. J Geriatr Cardiol. 2012 Jun;9(2):197-208. doi: 10.3724/SP.J.1263.2011.12221. PMID 22916068
- [Background] Wittchen HU, Jacobi F, Rehm J, Gustavsson A, Svensson M, Jonsson B, Olesen J, Allgulander C, Alonso J, Faravelli C, Fratiglioni L, Jennum P, Lieb R, Maercker A, van Os J, Preisig M, Salvador-Carulla L, Simon R, Steinhausen HC. The size and burden of mental disorders and other disorders of the brain in Europe 2010. Eur Neuropsychopharmacol. 2011 Sep;21(9):655-79. doi: 10.1016/j.euroneuro.2011.07.018. PMID 21896369
- See also: SNF-Grant — https://data.snf.ch/grants/grant/215033